CLINICAL TRIAL: NCT01975233
Title: WEB French Observatory
Brief Title: WEB French Observatory of the WEB Aneurysm Embolization System
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12001
Record Dates: First submitted 2013-10-25; First posted 2013-11-04 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Brain Aneurysm
Keywords: Endovascular; Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WEB Aneurysm Embolization System: Subjects aged ≥ 18 years, but ≤ 75 years requiring treatment for intracranial aneurysms.
  Interventions: Device: WEB Aneurysm Embolization System

INTERVENTIONS:
Device: WEB Aneurysm Embolization System — WEB Aneurysm Embolization System

SUMMARY:
An observational post-market, open label, multicenter Observatory. The decision to use a WEB device to treat the patients has been made before and independently of the decision to include the patient in the French Observatory.

DETAILED DESCRIPTION:
Subjects will be screened for Observatory eligibility after giving informed consent. The embolization procedure will be performed in the digital angiographic suite using standard angiographic techniques.

Initial analysis of Observatory data will be performed at completion of 12 month follow-up for the first thirty-five (35) subjects.

Subjects will be followed per Institution's standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The decision to use a WEB device to treat the patients has been made before and independently of the decision to include the patient in the French Observatory
2. Subject must be ≥ 18 years of age;
3. Subject must have an intracranial aneurysm requiring treatment according to a multidisciplinary decision. If the subject has an additional aneurysm requiring treatment, the additional aneurysm must not require treatment within 30 days of the index procedure;
4. Aneurysm to be treated must have the following characteristics:

   i. Morphology - saccular ii. Location:
   * Basilar apex (BA), or
   * Middle cerebral artery (MCA) bifurcation, or
   * Internal carotid artery (ICA) terminus
   * Anterior communicating artery (ACom)
   * Anterior cerebral Artery (ACA) iii. Diameter and width of the aneurysm is appropriate size for treatment with the WEB Aneurysm Embolization System per device Instructions for Use iv. Dome-to-Neck (DN) ratio ≥ 1.0
5. Subject must be considered by the physician to be available for subsequent visits;
6. Subject must be able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule;
7. Subject must sign and date CPP and/or CCTIRS/CNIL approved written informed consent prior to initiation of any clinical evaluation procedures, including screening procedures (if unable to sign for self, legal representative may do so where applicable).

Additional inclusion criterion for ruptured aneurysms:

For subjects with ruptured aneurysm: subject has ruptured aneurysm with Hunt & Hess Score of I, II, or III

Exclusion Criteria:

* 1. Subject is greater than 75 years of age; 2. Subject has more than one aneurysm requiring treatment within 30 days of index procedure; 3. Subject is female and pregnant or breast-feeding; 4. Subject has a known coagulopathy; 5. Subject has a known hemoglobinopathy or thrombocytopathy; 6. Subject has lesion with characteristics unsuitable for endovascular treatment; 7. Subject has vessel, tortuosity or morphology which could preclude safe access and support during treatment with clinical evaluation device; 8. Subject exhibits ischemic symptoms such as transient ischemic attacks, minor strokes, stroke-in-evolution within 30 days prior to enrollment; 9. Subject exhibits clinical or angiographic evidence of vasospasm; 10. Subject has physical, neurologic or psychiatric conditions, which preclude Subject's ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule; 11. Subject has known hypersensitivity to any component of the clinical evaluation device, procedural materials, or medications commonly used during the procedure; 12. Subject has received any investigational device for treatment of the target intracranial aneurysm prior to entry into this trial; 13. Subject has an acute life-threatening illness other than the neurological disease to be treated in this trial; 14. Subject has a life expectancy of less than 2 years due to other illness or condition (in addition to an intracranial aneurysm);

Additional Exclusion Criteria for unruptured aneurysms:

15. Subject has Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of subarachnoid/intracranial hemorrhage on presentation; 16. Subject has any circulatory, neurovascular, or cardiovascular medical conditions that have resulted in neurological symptoms;

Additional Exclusion Criteria for ruptured aneurysms:

17. Subject has a ruptured aneurysm and Hunt & Hess Score of IV or V;

Additional Imaging Exclusion Criteria:

18. Subject has CT or MRI evidence of intracranial tumor (except small meningioma) or any other intracranial vascular malformations on presentation; 19. Subject has angiographic evidence of vasculitis; 20. Microcatheter could not reach Subject's aneurysm to allow necessary access to treat with clinical evaluation device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The decision to use a WEB device to treat the patients has been made before and independently of the decision to include the patient in the French Observatory
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Durability of aneurysm occlusion | 12 months
  The following efficacy assessments will be performed to assess the efficacy of the WEB Aneurysm Embolization System in the endovascular treatment of aneurysms.
  1. Durability of occlusion compared to post-procedure imaging
  Durability is defined as:
  i. No worsening of Raymond Class from post-procedure result to follow-up result and ii. Not classified as "Recanalized"

SECONDARY OUTCOMES:
Recurrence/recanalization rate | 12 months
  Rate of aneurysm recanalization

OTHER OUTCOMES:
Modified Raymond Scale | 12 months
Percentage occlusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pierot, MD PhD, Principal Investigator — CHU REIMS
Locations (10):
- France (10):
  - CHU Pellegrin, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU Beaujon, Clichy
  - Hôpital Neurologique Pierre Wertheimer, Lyon
  - Hôpital Nord Laennec, Nantes
  - CHU La Miletrie, Potiers
  - CHU Reims - Hôpital Maison-Blanche, Reims
  - CHU Pontchailloux, Rennes
  - CHU Purpan, Toulouse
  - CHU Bretonneau, Tours

REFERENCES:
- See also: Clinical and Anatomical Follow-up in Patients With Aneurysms Treated With the WEB Device: 1-Year Follow-up Report in the Cumulated Population of 2 Prospective, Multicenter Series (WEBCAST and French Observatory). — http://www.ncbi.nlm.nih.gov/pubmed/26552042
- See also: WEB Treatment of Intracranial Aneurysms: Clinical and Anatomic Results in the French Observatory. — http://www.ncbi.nlm.nih.gov/pubmed/26514608
- See also: WEB Treatment of Intracranial Aneurysms: Feasibility, Complications, and 1-Month Safety Results with the WEB DL and WEB SL/SLS in the French Observatory. — http://www.ncbi.nlm.nih.gov/pubmed/25655876
- See also: Aneurysm Treatment With Woven EndoBridge in the Cumulative Population of Three Prospective Multicenter Series: 2-Year Follow-up — http://www.ncbi.nlm.nih.gov/pubmed/31960052